CLINICAL TRIAL: NCT05981625
Title: Desensitizing Effect and Tooth Color Change After Using Giomer-based Varnish Versus Bioactive Glass Air Polishing in Treating Cervical Hypersensitive Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, omnia samy Garouda, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14422022559057
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Dentin Hypersensitivity, Non-carious Cervical Lesions, Bioactive Glass Air Polishing, S-PRG
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Giomer varnish containing surface pre-reacted glass fillers (Experimental): Giomer-based varnish is a light-curable varnish/desensitizer. The surface pre-reacted glass (S-PRG) filler is a bioactive trilaminar structure with a multifunctional glass core embedded in resin matrix. It can release and recharge fluoride ions. When it becomes in contact with the oral fluids, it starts to bind to the collagen fiber and release six different types of ions like fluoride, calcium, phosphate that help in the formation of apatite crystals and seal the open dentinal tubules with a long-lasting effect Brand name: S_PRG (Shofu-Japan)
  Interventions: Other: Giomer varnish containing surface pre-reacted glass fillers
- Bioactive Glass Air Polishing (Active Comparator): Bioactive glass powder delivered by standalone air polishing system, is a bioactive material that reacts with saliva to deposit Hydroxycarbonate Apatite crystals (HCA), which is very strong and resilient. The continuous release of calcium ions promotes constant protection and long lasting seal of the tubules. Using the air polishing delivery system helps to provide a huge amount of calcium and phosphate particles at the exposed surface of the tooth. Moreover, the air pressure aids in pushing these particles inside the dentinal tubules to a considerable depth. Air polishing using such powder provides a bifunctional advantage of occluding the dentinal tubules. However, there is limited clinical trials testing the efficacy of the bioactive glass powder air polishing system in minimizing the dentin hypersensitivity
  Interventions: Other: Giomer varnish containing surface pre-reacted glass fillers

INTERVENTIONS:
Other: Giomer varnish containing surface pre-reacted glass fillers — Giomer varnish (PRG barrier coat) will used as the intervention agent in this study. , Giomer is considered as a hybrid material between the resins modified glass ionomers and the composite resins. It is composed of 45% Sio2, 24.5% Na2O, 24.5% Ca O and 6% P2O5
  . The presence of sodium is very important due to its bioactivity while the phosphate is responsible for the degree of degradation and formation of apatite. Based on this composition, giomer has several clinical applications in implant, periodontics, bone generation, pulp capping, Root canal treatment, as restorative materials, in air abrasion, enamel remineralization and finally dentin hypersensitivity

SUMMARY:
This trial is test the dentin hypersenstivity using Giomer based Varnish versus Bioactive glass air polishing system in patients with non-cervical lesions.

DETAILED DESCRIPTION:
To investigate the clinical effectiveness of Giomer based varnish versus Bioactive glass air polishing System in the management of dentin hypersensitivity and tooth color change in the cervical lesions.

P:Patient/Population: Middle aged patients complaining of cervical dentin hypersensitivity. I: Giomer varnish containing surface pre-reacted glass fillers. C: Bio-active glass air polishing system: O:Dentin Hypersenstivity (Primary Outcome) was assessed by three different stimuli (evaporative , thermal and tactile) . O: Color Change (Secondary Outcome). T: Baseline, T1, T2, T3. S:a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants complaining from dentin hypersensitivity.
* Middle aged patients.
* Good oral hygiene.

Exclusion Criteria:

* Pregnant women.
* Patients with allergy to any material used in this study.
* Smoking patients will affect the oral hygiene and periodontal health.
* Patients taking anti-inflammatory drugs that will affect the perception of hypersensitivity.
* Systemically compromised patients.
* Smokers.
* Patients received desensitization treatment in the last 6 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pain due to dentin hypersenstivity | baseline preoperative, immediate postoperative, 1 , 6 and 12-months' time
  Dentin hypersensitivity was assessed by three different stimuli (evaporative , thermal and tactile) to simulate the different situations in which Dentin hypersensitivity arises. Using the Visual Analog scale (VAS), the participant marks the pain intensity on a graduated 10 cm straight line (0
  = no pain, 10 = extreme pain)

SECONDARY OUTCOMES:
Color change (Tooth discoloration) | Baseline preoperative, immediate postoperative, 1,6 and 12-months time
  According to USPH criteria Alpha: Matches tooth Bravo: Acceptable mismatch Charlie: Unacceptable mismatch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravishankar P, Viswanath V, Archana D, Keerthi V, Dhanapal S, Lavanya Priya KP. The effect of three desensitizing agents on dentin hypersensitivity: A randomized, split-mouth clinical trial. Indian J Dent Res. 2018 Jan-Feb;29(1):51-55. doi: 10.4103/ijdr.IJDR_458_17. PMID 29442087
- [Background] West N, Seong J, Davies M. Dentine hypersensitivity. Monogr Oral Sci. 2014;25:108-22. doi: 10.1159/000360749. Epub 2014 Jun 26. PMID 24993261
- [Background] Favaro Zeola L, Soares PV, Cunha-Cruz J. Prevalence of dentin hypersensitivity: Systematic review and meta-analysis. J Dent. 2019 Feb;81:1-6. doi: 10.1016/j.jdent.2018.12.015. Epub 2019 Jan 11. PMID 30639724
- [Background] Freitas Sda S, Sousa LL, Moita Neto JM, Mendes RF, Prado RR. Dentin hypersensitivity treatment of non-carious cervical lesions - a single-blind, split-mouth study. Braz Oral Res. 2015;29:45. doi: 10.1590/1807-3107BOR-2015.vol29.0045. Epub 2015 Mar 10. PMID 25760065